CLINICAL TRIAL: NCT01161459
Title: Research Institute of Nephrology, Jinling Hospital
Brief Title: Treatment of Idiopathic Membranous Nephropathy With Tripterygium Wilfordii Plus Steroid vs Tacrolimus Plus Steroid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhi-Hong Liu, M.D. (Other)
Responsible Party: Sponsor-Investigator, Zhi-Hong Liu, M.D., professor, Nanjing University School of Medicine
Organization: Nanjing University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-1004
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Idiopathic Membranous Nephropathy
Keywords: Idiopathic Membranous Nephropathy; Treatment; FK506; Tripterygium wilfordii
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Tacrolimus; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tripterygium wilfordii (Experimental): 120mg/d for 6 months,then decrease to 60mg/d by 30mg/d every month for 12 months
  Interventions: Drug: Tripterygium wilfordii
- FK506 (Active Comparator)
  Interventions: Drug: FK506

INTERVENTIONS:
Drug: Tripterygium wilfordii — Tripterygium wilfordii 120mg/d Prednisone 30mg/d
  Other Names: TW
  Arms: Tripterygium wilfordii
Drug: FK506 — capsule
  Other Names: Tacrolimus + Prednisone 30mg/d
  Arms: FK506

SUMMARY:
The purpose of this study is: To explore the potential role of Tripterygium wilfordii plus steroid in the treatment of membranous nephropathy.

To investigate the safety and tolerability of Tripterygium wilfordii plus steroid

DETAILED DESCRIPTION:
Idiopathic membranous nephropathy is the most common cause of nephrotic syndrome in adults. Over the past decade, a number of studies have reported therapeutic efficacy for treatment with tacrolimus plus steroid in patients with nephrotic syndrome including patients with membranous nephropathy. This study will evaluate the safety and effectiveness of a traditional herbal extraction, Tripterygium wilfordii, plus steroid in reducing the amount of protein in the urine in patients with membranous nephropathy. A hundred patients with biopsy-proven membranous nephropathy will be recruited. They will be screened with a medical history, physical examination, blood tests, and an examination for infection, cancers, and other conditions that can cause membranous nephropathy. The investigators plan to conduct an open-label study of the efficacy and safety of Tripterygium wilfordii in the treatment of membranous nephropathy. Half of them will be treated with oral Tripterygium wilfordii plus steroids for 6 months, followed by 6 months of maintenance, and the other half treated with tacrolimus plus steroid as positive contrast. Proteinuria, renal function will be monitored. Complete remission is defined as 24-hour urinary protein excretion to less than 0.4 mg/day and serum albumin>35g/L. This study will explore the potential role of Tripterygium wilfordii in the treatment of membranous nephropathy, it's cost less .

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven idiopathic membranous nephropathy
2. Nephrotic syndrome with proteinuria ( > 3.5 g/day) and serum albumin < 30 g/dl
3. Age 18-65 years with informed consent

Exclusion Criteria:

1. Patient with elevated serum creatinine concentration
2. Prior therapy with sirolimus, CSA, MMF, or azathioprin, cytoxan, chlorambucil, levamisole, methotrexate, or nitrogen mustard in the last 90 days
3. Active/serious infection
4. Patient with hepatitis B surface antigen or who is hepatitis C antibody positive
5. Patient who is diabetic
6. Patient is allergic or intolerant to macrolide antibiotics or tacrolimus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The number of CR and PR of Tripterygium wilfordii plus steroid in the treatment of membranous nephropathy | 18 months

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerabilitysteroid | 18 months
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, Master, Principal Investigator — Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine
Locations (1):
- Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China